CLINICAL TRIAL: NCT07020195
Title: QFR-Based Functional SYNTAX Score System in Optimizing Revascularization Strategy for Multivessel Disease: A Prospective Multicenter Randomized Controlled Trial
Brief Title: QFR-Based Functional SYNTAX Score System in Optimizing Revascularization Strategy for Multivessel Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: QFR-FSS
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
Keywords: Multivessel Disease; QFR-Based Functional SYNTAX Score System
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional SYNTAX scoring (SS) (Active Comparator): Using traditional SYNTAX scoring to guide the selection of revascularization strategies
  Interventions: Procedure: Traditional SYNTAX scoring
- QFR-Based Functional SYNTAX Score System (QFR-FSS) (Experimental): Using QFR-Based Functional SYNTAX Score System to guide the selection of revascularization strategies
  Interventions: Procedure: QFR-Based Functional SYNTAX Score System

INTERVENTIONS:
Procedure: Traditional SYNTAX scoring — Using traditional SYNTAX scoring to guide the selection of revascularization strategies
  Arms: Traditional SYNTAX scoring (SS)
Procedure: QFR-Based Functional SYNTAX Score System — Using QFR-Based Functional SYNTAX Score System to guide the selection of revascularization strategies
  Arms: QFR-Based Functional SYNTAX Score System (QFR-FSS)

SUMMARY:
The revascularization treatment of multi vessel coronary artery disease (MVD) has always been a complex and important field in the treatment of coronary heart disease. The relative benefits of PCI and CABG vascular reconstruction strategies have always been a controversial topic in the field of MVD treatment. At present, SYNTAX score is the most commonly used imaging scoring system in clinical practice for quantitatively evaluating the complexity of coronary artery MVD, preliminary selection of revascularization strategies, and risk stratification. However, the SYNTAX score is entirely based on anatomical information of the lesion, and the assessment of the degree of coronary artery ischemia caused by the lesion is not accurate enough. Relying solely on anatomical structures for scoring may overestimate the harm of non ischemic lesions. The functional SYNTAX score (FSS) combines functional assessment of coronary artery lesions with anatomical structure scoring, only including lesions with hemodynamic significance, effectively optimizing the traditional SYNTAX scoring system. Compared with traditional SYNTAX scoring, FSS can reduce the number of high-risk patients, objectively evaluate the functional significance of lesions, and guide PCI treatment, significantly improving clinical prognosis.

Quantitative flow ratio (QFR) is a novel method for evaluating the functional significance of coronary artery stenosis. However, it is currently unclear whether FSS based on QFR can achieve objective and accurate risk stratification, guide the selection of revascularization strategies, and improve the long-term prognosis of patients with coronary artery MVD. Higher quality prospective clinical trials need to be designed for verification.

Therefore, this study will use a functional SYNTAX scoring system based on QFR (QFR-FSS) to conduct a prospective, multicenter, randomized controlled clinical trial to evaluate the guiding value of QFR-FSS in selecting revascularization strategies for patients with coronary artery MVD and its impact on long-term cardiovascular prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Diagnosed as MVD patient by coronary angiography (≥ 50% stenosis in ≥ 2 major vessels);
* Plan to undergo PCI or CABG treatment, and ensure that the contrast images meet the imaging quality requirements for QFR analysis;
* Voluntarily sign the informed consent form, be able to participate in randomization and cooperate in completing all follow-up visits.

Exclusion Criteria:

* Acute myocardial infarction requires emergency PCI;
* Severe left ventricular dysfunction (LVEF<30%) or cardiogenic shock;
* The quality of coronary angiography images is poor, such as vascular overlap, respiratory artifacts, projection angles less than 25 °, or frame rates less than 15 frames per second;
* Failure of QFR analysis due to severe calcified lesions (determined by the central laboratory);
* eGFR<30 mL/min/1.73m ² or contrast agent allergy;
* Patients using intravenous pressors, intra aortic balloon counterpulsation, or other mechanical circulatory support devices;
* Patients undergoing tracheal intubation treatment;
* Patients who have received thrombolytic therapy before admission;
* Pregnant women;
* Expected survival time<1 year due to non cardiac reasons;
* Patients who are not expected to receive antiplatelet therapy for at least 6 months;
* Patients who have received CABG treatment in the past or plan to receive CABG treatment;
* Patients who plan to undergo any surgical procedure within 6 months;
* There are other conditions that may interfere with follow-up, such as dementia, drug abuse including drug use and drug dependence for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of major adverse cardiovascular events (MACE) | 2 years
  The incidence of major adverse cardiovascular events (MACE) 2 years after PCI or CABG surgery, defined as the composite endpoint of all-cause mortality, myocardial infarction, and ischemia driven revascularization.

SECONDARY OUTCOMES:
Composite endpoint of cardiogenic death and myocardial infarction | 2 years
  Composite endpoint of cardiogenic death and myocardial infarction
Disease success rate | 2 years
  Disease success rate: including lesion success evaluated by contrast imaging (evaluated by the central laboratory, with a visual residual stenosis degree of less than 30% and TIMI blood flow grade 3 for lesions treated with stent implantation); The residual stenosis degree of lesions treated with balloon dilation is less than 50% visually, TIMI blood flow grade 3, and the functional evaluation of lesions is successful (evaluated by the central laboratory, QFR ≥ 0.80 immediately after surgery).
Clinical success rate | 2 years
  Clinical success rate: On the basis of successful imaging lesions at 30 days, 1 month, 6 months, 1 year, and 2 years after surgery, the incidence of MACE within the same hospitalization period (up to 7 days).
The incidence of myocardial infarction | 2 years
  The incidence of myocardial infarction at 30 days, 1 month, 6 months, 1 year, and 2 years after surgery, including perioperative myocardial infarction (SCAI definition) and spontaneous myocardial infarction.
The incidence of all revascularization | 2 years
  The incidence of all revascularization (ischemia driven, non ischemia driven revascularization; infarct related artery, non infarct related artery revascularization, culprit and non culprit lesion revascularization) at 30 days, 1 month, 6 months, 1 year, and 2 years after surgery.
The incidence of confirmed and possible stent thrombosis | 2 year
  The incidence of confirmed and possible stent thrombosis (ARC-2 definition) at 30 days, 1 month, 6 months, 1 year, and 2 years after surgery (including stent thrombosis within the time range of acute, subacute, late, and late onset).
Postoperative quality of life scores | 2 year
  Postoperative quality of life scores at 2 years (EQ-5D Scale).